CLINICAL TRIAL: NCT01975532
Title: Evaluation of MRI Based Fiber Tracking as a Tool in Deep Brain Stimulation for Movement Disorders
Brief Title: Evaluation of Diffusion MRI as a Tool in Planning Deep Brain Stimulation (DBS)
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 26-MRI-DTI-on-DBS
Record Dates: First submitted 2013-10-22; First posted 2013-11-04 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the relationship between deep brain stimulation implantation site and DTI (diffusion tensor imaging) derived measures for the region and later compare this to the clinical treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Deep Brian Stimulation surgery

Exclusion Criteria:

* DBS treatment stopped before 12 month followup

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients screened and deemed eligible for treatment with Deep Brain Stimulation
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
UPDRS (unified parkinson disease rating scale) score | patients will be followed from pre-surgical evaluation to 1 year after surgery, roughly 13-14 months

SECONDARY OUTCOMES:
Cognitive scores on neuropsychological exam | patients will be followed from per-surgical evaluation to 1 year after surgery, roughly 13-14 months

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Petersen, phd-student, Principal Investigator — Aarhus University Hospital